CLINICAL TRIAL: NCT05542498
Title: Mobile Mindfulness Training and Physics Learning
Brief Title: Promoting Stress Management and Engagement in Introductory Physics Courses with Mindfulness and Relaxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Galla, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19050258 Part 2
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Psychological Stress; Coping Skills; Emotions; Emotion Regulation
Keywords: Mindfulness; Physics Education; Psychological Challenge and Threat; Engagement; Motivation; Relaxation
MeSH Terms: conditions — Stress, Psychological; Emotional Regulation | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Training (Active Comparator): 5-lesson audio-guided mindfulness training program delivered over 5 consecutive days, with two additional writing activities on day 1 and day 5
  Interventions: Behavioral: Mindfulness
- Relaxation Training (Active Comparator): 5-lesson audio-guided relaxation training program delivered over 5 consecutive days, with two additional writing activities on day 1 and day 5
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Mindfulness — Training is focused on learning and applying the principles of R.A.I.N. (Recognize, Allow, Investigate, Non-identify) in the context of physics learning.
  Arms: Mindfulness Training
Behavioral: Relaxation — Training is focused on learning and applying relaxation practices (e.g., progressive muscle relaxation, guided imagery) in the context of physics learning.
  Arms: Relaxation Training

SUMMARY:
This study tests the impact of mindfulness vs. relaxation training on psychological threat and challenge, emotions/emotion regulation, motivation/engagement, and performance among undergraduates enrolled in introductory physics courses. Data used to compare groups will be collected from a variety of sources, including self-report surveys, experience sampling and daily diary assessments, physics learning activities, and academic records.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* current University of Pittsburgh undergraduate
* enrolled in introductory physics
* self-reports psychological threat in physics

Exclusion Criteria:

* under 18 years of age
* not a current University of Pittsburgh undergraduate
* not enrolled in introductory physics
* does not self-report psychological threat in physics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Change in Daily Physics Emotions from baseline up to 1 week post-intervention assessed via Daily Diary Self-Report | From enrollment up to 1 week post-intervention
  Daily Physics Emotions measured using 12 self-report items with Likert scale from 0 (not at all) to 4 (an extreme amount). Daily Physics Emotions are calculated by averaging daily emotion items, with scores closer to 4 indicating experiencing more extreme emotions in physics.
Mean Change in Daily Responses to Physics Emotions from baseline up to 1 week post-intervention assessed via Daily Diary Self-Report | From enrollment up to 1 week post-intervention
  Daily reappraisal, perspective shifting, and relaxation measured using 6 self-report items with Likert scale from 0 (not at all true) to 4 (completely true). Composite scores for reappraisal, perspective shifting, and relaxation are calculated as an average of all items for each subscale, respectively. Daily responses to emotions ranges from 0 to 4, with higher scores indicating greater use of reappraisal, perspective shifting, or relaxation.
Mean Change in Daily Threat vs. Challenge Appraisals from baseline up to 1 week post-intervention assessed via Daily Diary Self-Report | From enrollment up to 1 week post-intervention
  Daily Threat vs. Challenge Appraisals measured using 3 self-report items about threat, challenge, and confidence with regarding to unpleasant physics emotions with Likert scale from 1 (strongly disagree) to 6 (strongly agree).
Mean Change in Daily Physics Engagement from baseline up to 1 week post-intervention assessed via Daily Diary Self-Report | From enrollment up to 1 week post-intervention
  Degree to which students felt engaged in and motivated to learn physics on a daily basis. Measured using 2 self-report items measured with Likert scale from 1 (not at all motivated/engaged) to 6 (extremely motivated/engaged). Daily engagement is calculated by averaging both items, with scores closer to 6 indicating more greater physics engagement.

SECONDARY OUTCOMES:
State Presence assessed via Ecological Momentary Assessment | during intervention, five days
  Experiences of decentering and curiosity, measured using 6 self-report items with Likert scale from 0 (not at all) to 4 (very much). State presence is calculated by averaging decentering and curiosity items, with scores closer to 4 indicating greater state presence.
State Relaxation assessed via Ecological Momentary Assessment | during intervention, five days
  Experiences of relaxation, measured using 3 self-report items with Likert scale from 0 (not at all) to 4 (very much). State relaxation is calculated by averaging relaxation items, with scores closer to 4 indicating greater state relaxation.
State Physics Anxiety assessed via Ecological Momentary Assessment | during intervention, five days
  Current level of anxiety about physics measured using 1 self-report item with Likert scale from 0 (not at all) to 4 (very much), with scores closer to 4 indicating higher anxiety about physics.
Mean Change in Physics Anxiety from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Anxiety evaluation or learning while doing physics work, measured using 8 self-report items with Likert scale from 1 (low anxiety) to 5 (high anxiety). Physics anxiety is calculated as an average of all of the items for each subscale, respectively. Physics anxiety ranges from 1 to 5, with higher scores indicating greater physics anxiety.
Mean Change in Psychological Threat vs. Challenge from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Psychological Threat vs. Challenge, measured using 11 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Psychological threat is calculated by subtracting average of physics demands from average of physics resources. Difference score ranges from -5 to 5, with scores above zero indicating psychological threat and scores of 0 or lower indicating psychological challenge.
Mean Change in Unpleasant Emotions-Can-Be-Enhancing Mindset from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Belief that unpleasant emotions are a signal that learning and growth are possible, measured using 3 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Unpleasant Emotions-Can-Be-Enhancing mindset is calculated as an average of all items ranging from 1 to 6, with higher scores indicating greater endorsement of this mindset.
Mean Change in Physics Self-Efficacy from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Belief of efficacy with respect to physics skills and abilities, measured using 5 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Physics Self-Efficacy is calculated as an average of all items from 1 to 6, with higher scores indicating greater self-efficacy in physics.
Mean Change in Physics Belonging from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Student's sense of belonging in their physics course, measured using 5 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Physics Belonging is calculated as an average of all items from 1 to 6, with higher scores indicating greater sense of belonging in physics.
Mean Change in Metacognitive strategies from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Metacognitive strategies, measured using 7 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Metacognitive strategies are calculated as an average of all items, ranging from 1 to 6, with higher scores indicating greater use of metacognitive strategies.
Mean Change in Physics Intelligence Mindset from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Belief that intelligence and abilities for physics can be developed through dedication and hard work, measured using 3 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Growth mindset is calculated as an average of all items ranging from 1 to 6, with higher scores indicating greater growth mindset and lower scores indicating greater fixed mindset.
Mean Change in Cognitive Effort from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Cognitive effort, measured using 4 self-report items with Likert scale from (strongly disagree) to 6 (strongly agree). Cognitive effort is calculated as an average of all items, ranging from 1 to 6, with higher scores indicating greater cognitive effort.
Mean Change in Physics Identity from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  The degree by which students associate their self-concept with physics, measured using 4 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Physics Identity is calculated as an average of all items from 1 to 6, with higher scores indicating greater identification with physics.
Mean Change in Proactive Mindset from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Proactive mindset, measured using 6 self-report items with Likert scale from 1 (not at all) to 5 (very much). Proactive mindset is calculated as an average of all items, with higher scores indicating greater proactive mindset.
Mean Change in Cognitive Problem-Solving Strategies from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Use of explanation and analogy as problem solving strategies when working on physics, measured using 6 self-report items with Likert scale from (strongly disagree) to 6 (strongly agree). Each subscale is calculated as an average of all of the items for each subscale, respectively. Cognitive problem-solving strategies range from 1 to 6, with higher scores indicating greater use of explanation or analogy problem solving strategies.
Mean Change in Physics Value from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Perceived interest in and utility value of learning physics, measured using 2 self-report items with Likert scale from 1 to 6. Physics Value is calculated as an average of both items from 1 to 6, with higher scores indicating greater perceived value of learning physics.
Performance on Physics problem solving Tasks | 3 days post-intervention
  Physics problem solving tasks that range in difficulty covering content from introductory physics. Each item is scored for accuracy and solution time. Multiple choice items are scored as correct or incorrect. Accuracy scores are averaged across the items with higher scores indicating better physics performance.
Performance on the Preparation for Future Learning Task | 3 days post-intervention
  Physics problem solving tasks that include new learning resources (e.g., a worked example) and a transfer task. Each item is scored for accuracy and latency. Explanation items are scored on a rubric. Accuracy scores are summed across items with higher scores indicating better physics learning. Latencies will be examined for how much time was spent with the learning resource and time spent solving the problems.
Judgments of confidence, difficulty, and self-efficacy during the physics problem solving and Preparation for Future Learning tasks assessed via Self-Report | 3 days post-intervention
  Judgments of confidence, difficulty, and self-efficacy during physics problem solving, with each subscale measured using self-report items with Likert scale from 1 to 6. Each subscale is calculated as an average of all of the items, with higher scores indicating greater confidence, difficulty, and self-efficacy respectively.
Problem selection on a Make-a-Physics task | 3 days post-intervention
  Physics problem solving tasks that range in difficulty from more to less challenging. Participants select problems to be included on a work sheet. Scores are calculated by summing the number of problems selected for each problem type.

OTHER OUTCOMES:
Performance in Physics Class | End of semester following intervention, approximately 12 weeks
  End-of-course grades measured via school records. Higher grades indicate higher classroom performance.
Retention in Physics Classes | End of semester following intervention, approximately 7 months
  Enrollment in second semester of introductory physics course sequence measured via official school records. Scored dichotomously, 1 for enrolling second semester physics and 0 for not.
Mean Change in Mindfulness from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Trait decentering and curiosity, measured using 13 self-report items with Likert scale from 0 (not at all) to 5 (very much). Trait mindfulness is calculated as an average of all items, ranging from 0 to 5, with higher scores indicating greater mindful decentering and curiosity; will also be used as a covariate or moderator.
Mean Change in Rational-Experiential Ability from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  Trait rational-experiential ability, measured using 10 self-report items with Likert scale from 1 (strongly disagree) to 6 (strongly agree). Each subscale is calculated as an average of all of the items for each subscale, respectively. Higher scores indicate greater rational or experiential thinking abilities.
Mean Change in Knowledge Transfer from baseline up to 3 months post-intervention assessed via Self-Report | From enrollment, up to 3 months post-intervention
  General self-reported learning and transfer strategies, measured using 5 self-report items with Likert scale from (strongly disagree) to 6 (strongly agree). Physics Transfer is calculated as an average of all items, ranging from 1 to 6, with higher scores indicating greater use of learning and transfer strategies.
Treatment Expectancy assessed via Self-Report | 3 days post-intervention
  Perception of credibility and expected efficacy of training, measured using 4 self-report items with Likert scale from 1 (not at all) to 5 (very much). Each subscale is calculated as an average of all of the items for each subscale, respectively. Higher scores indicate greater perceived credibility or efficacy of the training.
Intervention Attention Check Questions assessed via Ecological Momentary Assessment | during intervention, five days
  Multiple choice questions gauging the attentiveness to the intervention audio. Each item is scored for accuracy, as correct or incorrect.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Galla, PhD, Principal Investigator — University of Pittsburgh; Timothy Nokes-Malach, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data and materials required to reproduce results reported in publications will be available to researchers.
Supporting Information: Analytic Code
Time Frame: Data, materials, and analytic code required to reproduce results will be shared upon publication.
Access Criteria: Data, materials, and analytic code will be shared on Open Science Framework (or other online repository).